CLINICAL TRIAL: NCT06753747
Title: A Phase 1b/2 Trial of Afatinib Plus Palbociclib in Previously Treated Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: A Trial of the Combination of Afatinib and Palbociclib in Previously Treated Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, professor, West China Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-143
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — palbociclib; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1b: Afatinib(30mg)+Palbociclib (Experimental): In phase 1b, there is 2 dose levels for Afatinib, 30mg qd and 40 mg qd, and if no patients experience DLT on 30mg level, 40mg level will be administered.
  Interventions: Drug: Palbociclib; Drug: Afatinib(30mg)
- Phase 1b: Afatinib(40mg)+Palbociclib (Experimental): In phase 1b, there is 2 dose levels for Afatinib, 30mg qd and 40 mg qd, and if no patients experience DLT on 30mg level, 40mg level will be administered.
  Interventions: Drug: Palbociclib; Drug: Afatinib(40mg)
- Phase 2: Afatinib(RP2D)+Palbociclib (Experimental): The RP2D of Afatinib determined in phase 1b will be administrated in phase 2
  Interventions: Drug: Palbociclib; Drug: Afatinib(RP2D)

INTERVENTIONS:
Drug: Palbociclib — Palbociclib will be given at a dose of 100 mg every day orally with three weeks on and one week off. Four weeks is a cycle.
Drug: Afatinib(30mg) — Afatinib will be administered orally at a dose of 30 mg once daily (QD) in each 4-week cycle.
  Arms: Phase 1b: Afatinib(30mg)+Palbociclib
Drug: Afatinib(40mg) — Afatinib will be administered orally at a dose of 40 mg once daily (QD) in each 4-week cycle.
  Arms: Phase 1b: Afatinib(40mg)+Palbociclib
Drug: Afatinib(RP2D) — In the Phase 2 study, the recommended Phase 2 dose (RP2D) of Afatinib, determined during the Phase 1b portion, will be utilized.
  Arms: Phase 2: Afatinib(RP2D)+Palbociclib

SUMMARY:
The goal of this clinical trial is to learn if Afatinib plus Palbociclib works in previously treated recurrent or metastatic esophageal squamous cell carcinoma. It will also learn about the safety of the combination of Afatinib and Palbociclib. The main questions it aims to answer are:

What is the safe and tolerable dose of Afatinib when combined with 100 mg of Palbociclib (administered orally, three weeks on and one week off)?

Does the combination therapy of Afatinib and Palbociclib induce a tumor response in patients with recurrent or metastatic esophageal squamous cell carcinoma who have received prior treatments?

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Histologically or cytologically confirmed as ESCC, locally advanced and unresectable, with local recurrence (local lymph node metastases) or distant metastases
* Immunohistochemistry confirmed EGFR(3+) or EGFR-FISH-amplification or next generation sequencing confirmed EGFR-amplification (EGFR expression is not required in Phase 1b, but only patients with EGFR overexpression will be included in Phase 2).
* Disease progression after first-line or subsequent lines of therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate organ function within 7 days prior to treatment initiation, meeting the following criteria:Hematology (without transfusion, blood products, or administration of G-CSF or other hematopoietic stimulants within the past 14 days):

  1. Hemoglobin (Hb) ≥ 90 g/L;
  2. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L;
  3. Platelet count (PLT) ≥ 75 × 10⁹/L.

Serum biochemistry:

1. Total bilirubin (TBIL) ≤ 1.5 × the upper limit of normal (ULN);
2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; for patients with liver metastases, ALT and AST ≤ 5 × ULN;
3. Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 60 mL/min. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%, as assessed by Doppler ultrasound.

Coagulation: International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN.

* Female patients of childbearing potential must agree to use appropriate contraception from screening until 3 months after the end of treatment and must not be breastfeeding. A negative pregnancy test is required within 7 days before the start of treatment. Male patients must agree to use appropriate contraception or have undergone surgical sterilization during the study and for 8 weeks after the last administration of study medication.
* All subjects are recruited on a voluntary basis and sign the informed consent. They are required to be compliant with the study and cooperative with the follow-up.

Exclusion Criteria:

* Patients who have a history of other malignancies in the past five years (except for the cured basal cell carcinoma and cervical carcinoma in situ)
* The patient has any active autoimmune disease or a history of autoimmune disease
* History of severe allergic reactions or known allergies to macromolecular protein preparations, Afatinib, Palbociclib, or any component of their formulations that have resulted in hospitalization.
* Presence of contraindications to Palbociclib or Afatinib.
* Previous or planned treatments as follows:

  1. Prior use of EGFR inhibitors or CDK4/6 inhibitors.
  2. Administration of any live vaccines (e.g., influenza or varicella vaccines) within 4 weeks before the first dose or during the study.
  3. Major surgery or significant trauma within 4 weeks before the first dose.
  4. Residual toxicities from prior anti-tumor therapies not resolved to ≤ Grade 1 per CTCAE v5.0, except for alopecia or platinum-based therapy-induced neuropathy.
* Severe medical conditions, such as:

  1. NYHA Class II or higher heart failure.
  2. Ischemic heart disease (e.g., myocardial infarction or angina).
  3. Clinically significant supraventricular or ventricular arrhythmias.
  4. Poorly controlled diabetes (fasting blood glucose ≥ 10 mmol/L).
  5. Poorly controlled hypertension (systolic BP > 150 mmHg and/or diastolic BP > 100 mmHg).
  6. Left ventricular ejection fraction (LVEF) < 50% on echocardiography.
  7. QTc interval > 450 ms in males or > 470 ms in females.
  8. Abnormal ECG findings deemed to pose additional risk by the investigator.
* Active infections or unexplained fever within 48 hours prior to the first dose, or systemic antibiotic use within one week prior to informed consent.
* Active hepatitis B (HBV DNA ≥ 2000 IU/mL or ≥ 10⁴ copies/mL), hepatitis C (anti-HCV antibody positive with detectable HCV RNA), known HIV positivity, or acquired immunodeficiency syndrome (AIDS).
* Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial.
* Pregnancy or lactation.
* Receipt of any investigational drug within 4 weeks before the first dose or concurrent enrollment in another clinical trial, except for observational (non-interventional) studies or interventional trials in follow-up.
* Any other factors deemed by the investigator to potentially interfere with study participation, including the ability to complete study treatment and follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Afatinib | from the first dose to within 30 days after the last dose
Objective Response Rate (ORR) | up to 2 years
  the proportion of patients with a confirmed complete response or partial response, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | from the first dose to within 30 days after the last dose
  Number of participants who experience grade 1 or higher adverse events, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)
Disease Control Rate (DCR) | up to 2 years
  Percentage of patients who achieve partial response (PR) or complete response (CR) or stable disease (SD) based on Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
Progression free survival | up to 2 years
  the time from treatment initiation to the first disease progression or death from any cause
Overall survival(OS) | up to 2 years
  the time from treatment initiation until death from any reason
Anti-tumor activity by Duration of Response (DOR) | up to 2 years
  Calculated as the average length of time between response to treatment and disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhou, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No